CLINICAL TRIAL: NCT05164510
Title: Exploratory Study on Gene Profiling of Circulating Tumor DNA（ctDNA） of Multiple Primary Cancers （MPC） and Its Value in Guidance of Clinical Choice of Drugs
Brief Title: Value of ctDNA in the Treatment of Multiple Primary Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan CMP-001
Record Dates: First submitted 2021-09-07; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-09

CONDITIONS: Multiple Primary Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ct-DNA test in MPC (Experimental): treatment according to ct-DNA results:For Patients with abnormal gene changes of corresponding targeted drugs are recommended to use corresponding targeted therapy or immunotherapy drugs;For Patients without abnormal gene changes of corresponding targeted drugs, Treatment of Physician's Choice (TPC) is recommended.
  Interventions: Genetic: ct-DNA guided therapy

INTERVENTIONS:
Genetic: ct-DNA guided therapy — treatment according to ct-DNA results:For Patients with abnormal gene changes of corresponding targeted drugs are recommended to use corresponding targeted therapy or immunotherapy drugs;For Patients without abnormal gene changes of corresponding targeted drugs, Treatment of Physician's Choice (TPC) is recommended.
  Other Names: treatment according to ct-DNA results

SUMMARY:
This trial is a single-center, prospective, exploratory study.The objective is to study the peripheral blood circulating tumor DNA (CT-DNA) gene profile of patients with multiple primary tumors (MPC) and to evaluate the exploratory study for guiding drug selection. Patients with multiple primary tumors who met the inclusion criteria and did not meet the exclusion criteria will be enrolled in this study. CtDNA test will be used for CT-DNA gene profile study, and whether the test results can guide drug selection will be evaluated.The expected enrollment time is 12 months, and clinical observation is performed until disease progression and patient death.Additional CT-DNA tests will be performed as the disease progresses (2 cT-DNA tests in total).

DETAILED DESCRIPTION:
This trial is a single-center, prospective, exploratory study.The objective is to study the peripheral blood CT-DNA gene profile of patients with multiple primary tumors and to evaluate the exploratory study for guiding drug selection. Patients with multiple primary tumors who met the inclusion criteria and did not meet the exclusion criteria will be enrolled in this study. CtDNA test will be used for CT-DNA gene profile study, and whether the test results can guide drug selection will be evaluated.The expected enrollment time is 12 months, and clinical observation is performed until disease progression and patient death. Additional CT-DNA tests will be performed as the disease progresses (2 cT-DNA tests in total).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were assessed to meet the diagnostic criteria for multiple primary tumors : each tumor had to be invasive histologically
* Each tumor has its own pathologic appearance
* Each tumor occurs in a different organ and must exclude metastasis or recurrence
* progress or failure after treatment on a standard regimen for related primary cancer
* regardless of gender, between 18 and 75
* The Eastern Cancer Collaboration Group (ECOG) scored 0 ~ 1 in physical condition (PS)
* has an estimated survival of more than three months;
* During 7 days (including 7 days) before screening, the laboratory test data were obtained: neutrophil count ≥1.5×109/L, platelet count ≥90×109/L, hemoglobin ≥90g/L (no transfusion within 14 days), serum total bilirubin ≤1.25 times normal upper limit (ULN);alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤ 2.5 x ULN (≤5x ULN in patients with liver metastasis);Serum creatinine ≤1.25 x ULN and creatinine clearance ≥60ml/min;
* Participating subjects (or their legal representative/guardian) had to sign an informed consent form saying they understood the study's objectives, understood the required procedures, and were willing to participate in the study.

Exclusion Criteria:

* have standard treatment for metastatic disease;
* Participants were given any experimental or antineoplastic drugs during the first four weeks of enrollment;
* Either symptomatic brain or meningeal metastasis (unless the patient is treated for something)At 6 months, imaging results were negative within 4 weeks prior to study entry and tumor-related clinical symptoms were stable at study entry);
* clinically active bleeding;
* Women who are pregnant or breastfeeding;Those who are fertile but do not take adequate contraceptive measures;
* addicted to alcohol or drugs;
* either major organ failure or other serious illness, including interstitial pneumonia, clinically relevant coronary disease, cardiovascular disease, or having myocardial infarction, congestive heart failure, unstable angina, pronounced pericardial effusion, or unstable arrhythmia in the first 6 months of the study;
* A history of severe neurological or mental illness;Severe infection;Active disseminated intravascular coagulation or other comorbidities that, in the investigator's judgment, seriously compromised the patient's safety or prevented the patient from completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
number of patients with aberrant CT-DNA gene profile | 8 months

SECONDARY OUTCOMES:
number of patients with drugable CT-DNA gene profile | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cencer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No